CLINICAL TRIAL: NCT07221331
Title: Prevalence, Clinical Characteristics, Progression, and Management of Neurofibromatosis Type 1 in Egypt (NF1-Egy)
Acronym: PRECIOUS Egypt
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D134BR00005
Record Dates: First submitted 2025-10-24; First posted 2025-10-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurofibromatosis type 1 (NF1), a genetic disorder, results from NF1 gene mutations with nearly complete penetrance (1). NF1 is considered common as a rare disease; it has a birth incidence of approximately one every 3000 and a prevalence of one case every 3000-6000 individuals.

Patients with NF1 present lifelong phenotypic variabilities, including those mentioned in the National Institutes of Health (NIH) diagnostic criteria: multiple cafe-au-lait macules, freckling, Lisch nodules, cutaneous neurofibromas, plexiform neurofibromas (PNs), optic pathway gliomas (OPG), and osseous lesions (1). Regarding PNs, they are present in about 30-50% of NF1 patients with deeper growth along internal nerve plexus cranial or large peripheral nerve sheaths, compared to cutaneous neurofibromas.

NF1 clinical expression is unpredictable, age-related, and varies among patients; additionally, as a tumor predisposition disorder, it is associated with neoplastic complications that impair health-related quality of life (QoL). Thus, it is essential to gather data about the natural history of the disease to understand its burden on patients with NF1 and those who develop PN.

Besides that, NF1 prevalence and patients' clinical characteristics are not well recognized in Egypt, and full surgical resection of PN is often challenging due to its invasive nature, location, and size. Accordingly, this is a disease registry to collect data about patients with NF1, both pediatrics and adults. And to understand the natural history of this disorder in Egypt over the past 14 years in real-world settings. For patients with NF1, with or without PNs, we aim to understand their treatment patterns and explore clinical and nonclinical factors influencing targeted outcomes.

ELIGIBILITY:
Inclusion Criteria:

A. Male or female patients of any age at index date (first diagnosis of NF1 and/or PN).

B. Have been diagnosed with NF1 according to the NIH Consensus Development Conference diagnostic criteria or the revised criteria between 01-Jan- 2010 and 31-December-2023.

Exclusion Criteria:

A. Missing NF1 diagnosis data in their medical record.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients' records will be eligible for study inclusion if the NF1 diagnosis date is between 01-Jan-2010 and 31-Dec-2023.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with Neurofibromatosis type 1-Plexiform Neurofibromas | 13 Years
  Prevalence of patients with NF1-PN from total NF1 population.

SECONDARY OUTCOMES:
Demographics | 13 Years
  Age at first diagnosis of NF1
Clinical characteristics | 13 Years
  Medical and surgical history
Patient management | 13 Years
  NF1-related medication history
Patient progression | 13 Years
  describe change in the growth of PN

CONTACTS AND LOCATIONS:
Locations (8):
- Egypt (8):
  - Research Site, Al Mansurah
  - Research Site, Alexandria
  - Research Site, Aswān
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, Sohag
  - Research Site, Tanta
  - Research Site, Zagazig

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/